CLINICAL TRIAL: NCT01217021
Title: An Exploratory, Open-label, Non-randomized Phase 0 Study to Evaluate Efficacy & Safety of MNI-558 Positron Emission Tomography for Detection/Exclusion of Cerebral Amyloid Beta in Patients w/ Alzheimer Disease Compared to Healthy Volunteers
Brief Title: Safety and Efficacy of Positron Emission Tomography (PET) Imaging With MNI-558
Acronym: MNI-558
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Danna Jennings, MD / Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-558-01
Record Dates: First submitted 2010-10-01; First posted 2010-10-08 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [18F] MNI-558 and PET imaging (Experimental)
  Interventions: Drug: [18F] MNI-558

INTERVENTIONS:
Drug: [18F] MNI-558 — Subjects will be injected with 5mCi, not to exceed >10% of 5mCI, of [18F]MNI-558, followed by PET imaging.

SUMMARY:
This research will look at how the brain may change in people with Alzheimer disease (AD).

The purpose of this research is to find out whether changes in the brain in people with Alzheimer disease can be detected using a brain imaging test. Most people with Alzheimer disease have changes in the brain that result in deposits of a protein called beta-amyloid. In this study, the investigators will be using a radioactive drug, [18F]MNI-558 that binds to beta-amyloid. This drug is experimental and has not been approved by the FDA. Brain imaging using PET (positron emission tomography) will be done to see if the investigators can evaluate the areas of beta-amyloid in the subjects with Alzheimer disease. The investigators will compare these scans with those done in healthy normal volunteers. PET is a brain-scanning test used in medicine and scientific research to see how the brain is working. The PET imaging test used in this study is not being done for diagnostic purposes.

DETAILED DESCRIPTION:
This is a phase 0, open-label, single-center, non-randomized single dose study to assess the safety and efficacy of MNI-558 PET imaging in detecting amyloid beta plaque in the brain in patients with probable AD compared to HVs. All aspects related to image acquisition, processing and visual as well as quantitative evaluation will be developed, optimized and validated (where required).

Each subject will be required to visit the study center during the screening phase, on the MNI-558 PET imaging day (baseline), and for 1 follow-up visit on the next day. A telephone follow-up visit will be performed 7 days after MNI-558 PET administration.

At the screening visit, each subject and the caregiver will be asked to provide written informed consent or assent. During the screening phase (maximum duration - 28 days) subject medical, neurological and surgical history, clinical assessments and a neuro-psychiatric evaluation will be performed on all eligible subjects. Subjects will be allowed to leave the center after all evaluations have been completed. During this period an MRI of the brain must be performed. During the MNI-558 PET imaging day, all subjects will receive a single IV injection of IMP and scanning will be performed from 0-60 min, 75-135 min, and 150-210 min (p.i). Each subject will be asked to return to the site for a follow-up visit (20 to 28 hours after IMP administration) and a telephone follow-up will occur 7 days thereafter. Safety will be assessed during both follow-up visits.

ELIGIBILITY:
Inclusion Criteria: ALL PARTICIPANTS

* is a man or woman and is ≥ 55 of age, whereby females must be without childbearing potential (confirmed by either: age ≥ 60; or history of surgical sterilization or of hysterectomy, or last spontaneous bleeding at least 2 years prior to the study start)
* has at least 6 years of education
* is able to provide informed consent or assent, and exhibits adequate visual, auditory and communication capabilities to enable compliance with study procedures. This includes performing the psychometric testing and being able to lie down flat in the PET scanner
* possesses a general health that permits adequate compliance with all study procedures as ascertained by a detailed review of the medical history, laboratory and physical examination findings, which must be performed within 28 days prior to administration of IMP
* the subject, or the subject and caregiver (for probable AD patients) will be compliant and have a high probability of completing the study in the opinion of the investigator
* informed consent has been signed and dated (with time) by the subject and/or the subject's caregiver (for probable AD patients)

Exclusion Criteria: ALL PARTICIPANTS

* has any contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan
* is scheduled for surgery and/or another invasive procedure within the time period of up to 24 hours following IMP application
* is allergic to the IMP or any of its constituents and/or has a history of severe allergic reactions to drugs or allergens (e.g. patients / volunteers with allergic asthma)
* is critically ill and/or medically unstable and whose clinical course during the observation period is unpredictable, e.g. patients / volunteers within 14 days of myocardial infarction or stroke, unstable patients / volunteers with previous surgery (within 7 days), patients with advanced heart insufficiency (NYHA stage IV), or with acute renal failure
* has a history of exposure to any radiation >15 mSv/year (e.g. occupational or radiation therapy)
* is receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g. chemotherapy)
* has received anti-amyloid drug therapy.
* has received any contrast material (X-ray, MRI) or radiopharmaceuticals within 48 hours prior to the application of the IMP or for whom application of such a substance is planned for the 24 hours following IMP administration
* has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening, and/or any radiopharmaceutical within 10 radioactive half-lives prior to IMP administration
* has a brain tumor or other intracranial lesion, a disturbance of CSF circulation (e.g., normal pressure hydrocephalus) and/or a history of head trauma or brain surgery
* has an inflammatory or infectious CNS disease, e.g. multiple sclerosis, HIV, syphilis, or Creutzfeld-Jacob disease
* has a history, physical, laboratory or imaging findings indicative of a significant neurological or psychiatric illness (for patients - other than AD)
* has another disease that can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function)
* has a history of alcohol or drug abuse
* has history of severe persistent depression

Inclusion Criteria: HEALTHY VOLUNTEERS

* has no evidence of cognitive impairment as indicated by a clinical dementia rating (CDR, [Hughes et al. 1993]) score of 0 (zero) and a score of ≥ 28 in the Mini-Mental Status Examination (MMSE, [Folstein et al. 1975])
* has in the CERAD neuropsychological test battery [Welsh et al. 1994] a z- score of ≥ (-1.00) for each subtest (except for the MMSE which is covered by criterion 1 above)
* has MRI brain scan that has been judged as "normal (age- appropriate)" including ARWMC scale [Wahlund et al. 2001] scores supporting the lack of cerebrovascular disease (e.g., a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1) and a Scheltens scale [Scheltens et al. 1992] verifying the lack of cerebral atrophy (e.g. bilateral temporal lobe atrophy visual score of 0 or 1)

Inclusion Criteria: ALZHEIMER DISEASE

* presents with positive assessment for dementia of Alzheimer's type in accordance with the DSM-IV-TR and probable AD according to the NINCDS-ADRDA criteria and fulfils none of the exclusion criteria of either (see Appendix 1,2)
* does not fulfill the ICC criteria for probable DLB (Appendix 3), the NINDS-AIREN for probable Vascular dementia (Appendix 5), or the Neary [Neary et al. 1998] criteria for FTD (Appendix 4)
* has a CDR [Hughes et al. 1993] score of 0.5, 1 or 2
* MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease (e.g., the ARWMC scale) changes limited to: a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1)
* has a caregiver who is willing and able to attend all study visits and perform the psychometric tests requiring the presence of a caregiver

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy safety of MNI-558 positron emission tomography (PET) for detection/exclusion of cerebral amyloid beta in patients with Alzheimer disease (AD) compared to healthy volunteers (HV) | 1 year
  To determine diagnostic efficacy of the MNI-558 PET scans in differentiating between patients with probable AD and HVs on the basis of neocortical tracer binding pattern, the PET scans will be visually assessed by a nuclear physician experienced in the field of neuro-imaging.
  Safety will be assessed from the rates of adverse events (AEs), changes in vital signs, changes in ECG parameters, changes in physical examination findings, changes in clinical laboratory findings, changes in injection site monitoring at pre-specified time points before and after IMP administration

SECONDARY OUTCOMES:
To assess the dynamic uptake of MNI-558, a potential imaging biomarker for B-amyloid burden in brain, using positron emission tomography (PET) in similarly aged Alzheimer (AD) subjects and healthy volunteers (HV | 1 year
  Images will be regionally analyzed by applying VOIs to the brain regions indicated above based on PET images coregistered with MRI images; SUV ratios and % injected dose concentrations will be determined using standardized image processing algorithms and commercial algorithms. Standard uptake values (SUV) are calculated for the areas of interest by using the established methods for normalizing to subject weight and injected dose.
To determine pharmacokinetics pattern of MNI-558 in venous plasma of healthy and AD subjects. | 1 year
  The concentration-time profile of total [F18]-radioactivity in plasma will be determined. The PK parameters Cmax, tmax and the AUC(0-tlast) (expressed in %ID*h/mL) of F-18-radioactivity will be derived from the concentration -time profile. The fraction of unchanged tracer in venous plasma at given time points will be determined by HPLC. The metabolite pattern will be described for each sampling time point. Blood sampling, radioactivity measurements of biological samples, generation of plasma samples, sample preparation and subsequent HPLC analyses will be done at the clinical study site.
To determine metabolite pattern of MNI-558 in venous plasma of healthy and AD subjects. | 1 year
  The concentration-time profile of total [F18]-radioactivity in plasma will be determined. The PK parameters Cmax, tmax and the AUC(0-tlast) (expressed in %ID*h/mL) of F-18-radioactivity will be derived from the concentration -time profile. The fraction of unchanged tracer in venous plasma at given time points will be determined by HPLC. The metabolite pattern will be described for each sampling time point. Blood sampling, radioactivity measurements of biological samples, generation of plasma samples, sample preparation and subsequent HPLC analyses will be done at the clinical study site.

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States